CLINICAL TRIAL: NCT06697392
Title: Ultrasound-based Artificial Intelligence for Grading of Carpal Tunnel Syndrome, a Multicenter Study in China
Brief Title: Ultrasound-based Artificial Intelligence for Classification of Carpal Tunnel Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Shi Xiaochen, Doctor, Peking University People's Hospital
Other Study IDs: 2024PHB019-001(5)
Record Dates: First submitted 2024-11-17; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Carpal Tunnel Syndrome (CTS); Ultrasound; Artificial Intelligence (AI)
Keywords: carpal tunnel syndrome; ultrasound; artificial intelligence
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prospective test set
  Interventions: Other: ultrasound examination

INTERVENTIONS:
Other: ultrasound examination — The investigators intend to perform ultrasound examinations for the participants with CTS.

SUMMARY:
Carpal tunnel syndrome (CTS) is one of the most prevalent peripheral neuropathies, impacting approximately 4% of the general population. It is typically classified into three degrees: mild, moderate, and severe. Accurate grading of carpal tunnel syndrome (CTS) is essential for determining appropriate treatment options, thereby playing a crucial role in optimizing patient outcomes. Electrophysiological testing (EST) is a key parameter for grading carpal tunnel syndrome (CTS). However, it is limited by several factors, including its invasive nature, poor reproducibility, and reduced sensitivity for detecting early-stage disease. Recently, ultrasound has gained widespread acceptance among clinicians for the assessment and grading of CTS. Nonetheless, radiologists often encounter challenges in this process due to the variability in image quality, differences in experience, and inherent subjectivity.

To address these issues, artificial intelligence presents a promising solution. Therefore, this study aims to develop a deep learning model for grading CTS by leveraging multimodal imaging features, including B-mode ultrasound, superb microvascular imaging (SMI), and elastography. Additionally, the investigators intend to validate the model's effectiveness by testing it with images from various clinical centers, ensuring its generalizability across different clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* those who have complained about associated symptoms about CTS, including pain, numbness, and weakness of hand.
* those who perform ultrasound examinations of median nerve within 1 week of the symptom.
* those who have electrophysilogical test results as reference standard.

Exclusion Criteria:

* those who had a surgery in the affected hand.
* those who had a trauma or fracture in the affected hand.
* those who had rheumatoid-related conditions, autoimmune diseases, and endocrine disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators intend to perform ultrasound examinations for patients with idiopathic CTS adhering to specific inclusion and exclusion criteria, aiming to develop and test the efficacy of AI model for CTS grading.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
grading of CTS | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing. PR, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chan HP, Samala RK, Hadjiiski LM, Zhou C. Deep Learning in Medical Image Analysis. Adv Exp Med Biol. 2020;1213:3-21. doi: 10.1007/978-3-030-33128-3_1. PMID 32030660
- [Background] Wielemborek PT, Kapica-Topczewska K, Pogorzelski R, Bartoszuk A, Kochanowicz J, Kulakowska A. Carpal tunnel syndrome conservative treatment: a literature review. Postep Psychiatr Neurol. 2022 Jun;31(2):85-94. doi: 10.5114/ppn.2022.116880. Epub 2022 May 31. PMID 37082094
- [Background] Lam KHS, Wu YT, Reeves KD, Galluccio F, Allam AE, Peng PWH. Ultrasound-Guided Interventions for Carpal Tunnel Syndrome: A Systematic Review and Meta-Analyses. Diagnostics (Basel). 2023 Mar 16;13(6):1138. doi: 10.3390/diagnostics13061138. PMID 36980446